CLINICAL TRIAL: NCT03148353
Title: Comparative Effectiveness of the Standardized and Modified Ultrasound Guided Corticosteroid Subacromial Injection for Participants With Shoulder Impingement Syndrome
Brief Title: Standardized and Modified Corticosteroid Subacromial Injection for Shoulder Impingement Syndrome
Acronym: SMCSINJ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201701028RIND
Record Dates: First submitted 2017-04-27; First posted 2017-05-11 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2017-05

CONDITIONS: Shoulder Impingement
Keywords: ultrasonography, corticosteroid, subacromial impingement syndrome, shoulder pain
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The treatment is double blind to the participants and outcome assessors. Only the physician performs the injection knows which kind of intervention the patients receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified subacromial injection (Experimental): 1. Intervention procedure: corticosteroid injection into the subacromial bursa and biceps tendon
     * Device for guidance: high-resolution ultrasound
     * Drug: 40 mg triamcinolone acetonide (a kind of corticosteroid)
  2. Intervention procedure: lidocaine injection into the subacromial bursa and biceps tendon
     * Device for guidance: high-resolution ultrasound
     * Drug: 3 mL of lidocaine (the medication will be mixed with 40 mg triamcinolone acetonide)
  Interventions: Procedure: Subacromial injection
- Standardized subacromial injection (Placebo Comparator): 1. Intervention procedure: corticoseroid injection into the subacromial bursa only
     * Device for guidance: high-resolution ultrasound
     * Drug: 40 mg triamcinolone acetonide (a kind of corticosteroid)
  2. Intervention procedure: lidocaine injection into the subacromial bursa only
     * Device for guidance: high-resolution ultrasound
     * Drug: 3 mL of lidocaine (the medication will be mixed with 40 mg triamcinolone acetonide)
  Interventions: Procedure: Subacromial injection

INTERVENTIONS:
Procedure: Subacromial injection — 1. Modified ultrasound guided corticosteroid subacromial injection
  2. Standardized ultrasound guided corticosteroid subacromial injection

SUMMARY:
Subacromial injection is a useful procedure to counteract shoulder impingement syndrome. With the aid of high-resolution ultrasound, the needle can be introduced precisely into the subacromial/subdeltoid bursa located between the acromion above and the supraspinatus tendon below. The standardized method allows the injectate to distribute along the subdeltoid bursa, further reliving pain from subacromial/subdeltoid impingement. In a substantial part of shoulder pain patients, it is common to accompany pain along the bicipital groove, which the biceps long head tendon courses through. The biceps long head tendon is attached to the superior labrum of the glenoid cavity and acts as the second important structure to prevent upward migration of the humeral head, following the supraspinatus tendon. Overuse injury of the biceps tendon is a likely cause of anterior shoulder pain. Concomitant administration of medication into the subacromial bursa and biceps tendon sheath is theoretically more effective than injection to the subacromial bursa only because the formal procedure targets two vulnerable structures in shoulder impingement syndrome at once. Regarding the standard ultrasound-guided subacromial injection. Therefore, we will conduct a randomized controlled trial investigating the effectiveness of standard subacromial injection in comparison with a novel approach simultaneously injecting the subacromial bursa and biceps tendon sheath.

DETAILED DESCRIPTION:
Introduction Subacromial injection is a useful procedure to counteract shoulder impingement syndrome. With the aid of high-resolution ultrasound, the needle can be introduced precisely into the subacromial/subdeltoid bursa located between the acromion above and the supraspinatus tendon below. The standardized method allows the injectate to distribute along the subdeltoid bursa, further reliving pain from subacromial/subdeltoid impingement. In a substantial part of shoulder pain patients, it is common to accompany pain along the bicipital groove, which the biceps long head tendon courses through. The biceps long head tendon is attached to the superior labrum of the glenoid cavity and acts as the second important structure to prevent upward migration of the humeral head, following the supraspinatus tendon. Overuse injury of the biceps tendon is a likely cause of anterior shoulder pain. Concomitant administration of medication into the subacromial bursa and biceps tendon sheath is theoretically more effective than injection to the subacromial bursa only because the formal procedure targets two vulnerable structures in shoulder impingement syndrome at once. Regarding the standard ultrasound-guided subacromial injection. Therefore, we will conduct a randomized controlled trial investigating the effectiveness of standard subacromial injection in comparison with a novel approach simultaneously injecting the subacromial bursa and biceps tendon sheath.

Material and methods:

Participants: adult patients (>20 year old) with shoulder impingement syndrome Inclusion criteria: shoulder pain>3 weeks; no contraindication for local injection; Visual analogue scale of pain>4 Participant number: at least 30 at each treatment arm Exclusion criteria: systemic rheumatologic disease, Ankylosing spondylitis, malignancy, major trauma or recent injections on the affected shoulder Study design: single center double blind randomized controlled trial Randomization method: block randomization (block size: 4), computerized random sequence generation, allocation concealment (+) Detail of the intervention

1. Control group: ultrasound guided injection into the subacromial bursa with 40 mg triamcinolone acetonide plus 3 mL of lidocaine
2. Experimental group: ultrasound guided injection into the subacromial bursa and biceps tendon sheath with 40 mg triamcinolone acetonide plus 3 mL of lidocaine

Outcome measurement:

Visual analogue scale of pain, physical examination(bicipital groove compression test, Speed's test, Yergason's test, empty can test, Neer's impingement test, Hawkins-Kennedy impingement test, painful arc test), range of motion, shoulder pain and disability index (SPADI), shoulder sonography (gray-scale/elastography)

Statistical analysis:

Continuous variables

1. Student's t test: fit assumption of normal distribution
2. Mann-Whitney test: does not fit the assumption of normal distribution Categorical variables

(1) Chi-square test (2) Fisher exact test: sparse data

Multivariate analysis:

1. Linear regression
2. Logistic regression Keywords: ultrasonography, corticosteroid, subacromial impingement syndrome, shoulder pain

ELIGIBILITY:
Inclusion Criteria:

* shoulder pain>3 weeks; no contraindication for local injection; Visual analogue scale of pain>4

Exclusion Criteria:

* systemic rheumatologic disease, Ankylosing spondylitis, malignancy, major trauma or recent injections on the affected shoulder

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Change in shoulder pain and disability index (SPADI) | Within 3 months after injection
  Shoulder pain and disability index (SPADI). The SPADI contains 13 items that assess two domains; a 5-item subscale that measures pain and an 8-item subscale that measures disability.

SECONDARY OUTCOMES:
Change in visual analogue scale of pain | within 3 months after injection
  The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be' . The patient is asked to mark his pain level on the line between the two endpoints.
Change in elasticity (strain ratio) | within 3 months after injection
  Change in tendon elasticity (strain ratio) after injection. Strain ratio is calculated for the target by selecting a region of interest (ROI) and a corresponding ROI of the adjacent reference tissue. Using machine inherent software, the strain ratio value is displayed on a static image.

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Vin Chang, MD, Principal Investigator — National Taiwan University Hospital Bei-Hu Branch
Locations (1):
- National Taiwan University Hospital, Bei-Hu branch, Taipei, Taiwan, Province of China, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chang KV, Wu WT, Han DS, Ozcakar L. Static and Dynamic Shoulder Imaging to Predict Initial Effectiveness and Recurrence After Ultrasound-Guided Subacromial Corticosteroid Injections. Arch Phys Med Rehabil. 2017 Oct;98(10):1984-1994. doi: 10.1016/j.apmr.2017.01.022. Epub 2017 Feb 27. PMID 28245972
- [Result] Cole BF, Peters KS, Hackett L, Murrell GA. Ultrasound-Guided Versus Blind Subacromial Corticosteroid Injections for Subacromial Impingement Syndrome: A Randomized, Double-Blind Clinical Trial. Am J Sports Med. 2016 Mar;44(3):702-7. doi: 10.1177/0363546515618653. Epub 2015 Dec 30. PMID 26717970
- [Derived] Hsu PC, Chang KV, Wu WT, Wang JC, Ozcakar L. Effects of Ultrasound-Guided Peritendinous and Intrabursal Corticosteroid Injections on Shoulder Tendon Elasticity: A Post Hoc Analysis of a Randomized Controlled Trial. Arch Phys Med Rehabil. 2021 May;102(5):905-913. doi: 10.1016/j.apmr.2020.11.011. Epub 2020 Dec 15. PMID 33338463
- [Derived] Wang JC, Chang KV, Wu WT, Han DS, Ozcakar L. Ultrasound-Guided Standard vs Dual-Target Subacromial Corticosteroid Injections for Shoulder Impingement Syndrome: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2019 Nov;100(11):2119-2128. doi: 10.1016/j.apmr.2019.04.016. Epub 2019 May 29. PMID 31150601
- See also: Static and Dynamic Shoulder Imaging to Predict Initial Effectiveness and Recurrence After Ultrasound-guided Subacromial Corticosteroid Injections. Archive of Physical Medicine and Rehabilitation. 2017 — http://www.ncbi.nlm.nih.gov/pubmed/28245972
- See also: Ultrasound-Guided Versus Blind Subacromial Corticosteroid Injections for Subacromial Impingement Syndrome: A Randomized, Double-Blind Clinical Trial. Am J Sports Med. 2016 — http://www.ncbi.nlm.nih.gov/pubmed/26717970